CLINICAL TRIAL: NCT02200731
Title: FAMOS: The Effect of Psychosocial Intervention for Childhood Cancer Survivors and Their Families: A Randomized Controlled Trial
Brief Title: FAMily Oriented Support (FAMOS): Psychosocial Intervention for Childhood Cancer Survivors and Their Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pernille Bidstrup (Other)
Collaborators: Rigshospitalet, Denmark (Other); Odense University Hospital (Other); Aarhus University Hospital Skejby (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Pernille Bidstrup, PhD, group leader, Danish Cancer Society
Organization: Danish Cancer Society (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FAMOS
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Childhood Cancer
Keywords: Childhood cancer; Psychosocial intervention; Family; Siblings; Childhood cancer survivors; Cogntive Behavioural; Manualized
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FAMOS: psychosocial family intervention (Experimental): The FAMOS intervention consists of a six session manualized psychosocial intervention including videos and tools. Four sessions focus on the parents and two sessions focus on the childhood cancer survivor and its siblings. The intervention is conducted by a psychologist with Cognitive Behavioral Therapy experience.
  Interventions: Behavioral: FAMOS: psychosocial family intervention
- Control (No Intervention): In Denmark, standard care after treatment does not include systematic psychosocial support. Families are able to seek support on their own or contact a support group offered by the Danish Cancer Society. However support specializing the families with childhood cancer survivors and their siblings after ending medial treatment is limited.

INTERVENTIONS:
Behavioral: FAMOS: psychosocial family intervention — The FAMOS intervention consists of a six session manualized psychosocial intervention including videos and tools. Four sessions focus on the parents and two sessions focus on the childhood cancer survivor and its siblings. The intervention is conducted by a psychologist with Cognitive Behavioral Therapy experience
  Arms: FAMOS: psychosocial family intervention

SUMMARY:
To investigate whether a home-based psychosocial family intervention that takes place shortly after ending the primary medical treatment can help families adjust to their cancer-related psychological issues.

DETAILED DESCRIPTION:
The objective of this randomized controlled trial is to investigate whether home-based psychosocial interventions are able to help families of childhood cancer survivors cope with cancer-related psychological issues.

Method: 300 families will be recruited from the four pediatric oncology departments in Denmark where 150 families' will receive a home-based psychosocial intervention and 150 families will be in the control group. The study will take place shortly after the child completes the primary treatment. The primary outcome is post-traumatic stress symptoms (PTSS) in parents and secondary outcomes include among others quality of life, sick-leave, coping strategies and family functioning. Families in the intervention group will receive a 6 session manualized intervention based on a Cognitive Behavioral framework. Four sessions will focus on the parents and two sessions will focus on the child, who had cancer, and his/her siblings. The main goal of the sessions is to teach families how to adapt healthy psychological adjustments to pediatric oncology and prevent PTSS in family members. As a part of the intervention, families will be presented with video clips of other parents discussing how cancer has affected their family, to show common issues in experiencing having a child undergo cancer treatment. Every family member will be asked to complete a set of questionnaires to measure the outcome of the intervention at baseline before the intervention, 6 months follow-up and 12 months follow-up.

It is expected that families in the intervention group experience a larger improvement in their post-traumatic stress symptoms as well as strengthening the family function, quality of life and reducing sick leave compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Families of children in the age range of 0-17 years diagnosed with any kind of cancer and treated at one of the four pediatric oncology departments in Denmark are invited to participate in the project after ending primary medical treatment.

Exclusion Criteria:

* If the child has a severe co-morbidity
* If the child has a mental disorder at diagnosis
* If the child is declared terminal ill at the end of treatment (less than 6 months of survival).
* If the parents and the children do not speak Danish. The participants have to be able to read and answer the questionnaires at the least, to be included in the project.
* If the parents do not wish to hand in consent form
* If the family participates in another randomized psychosocial intervention project

Max Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Post traumatic stress symptoms (PTSS) in parents measured by Harvard Trauma Questionnaire (HTQ) | Baseline and 6 months
  A larger reduction in post traumatic stress symptoms amongst parents of childhood cancer survivors in the intervention group from baseline to 6 months follow up compared to parents in the control group

SECONDARY OUTCOMES:
Post traumatic stress symptoms (PTSS) in parents measured by Harvard Trauma Questionnaire (HTQ) | Baseline and 12 months
  A larger reduction in post traumatic stress symptoms amongst parents of childhood cancer survivors in the intervention group from baseline to 12 months follow up versus parents in the control group
Post traumatic stress symptoms (PTSS) in childhood cancer survivors and their siblings measured by Harvard Trauma Questionnaire (HTQ), Daryl or Pediatric Emotional Distress Scale (PEDS) | Baseline, 6 months and 12 months
  A larger reduction in PTSS from baseline to respectively 6 and 12 months follow up in childhood cancer survivors and their siblings the intervention group versus the control group measured by Harvard Trauma Questionnaire (HTQ), Daryl or Pediatric Emotional Distress Scale (PEDS)
Family psychosocial functioning measured by Psychological Assessment Tool 2.0 (PAT2.0) and Family Impact Module 2.0 (FIM2.0) | Baseline, 6 months and 12 months
  An larger enhancement in the family's' psychosocial functioning from baseline to 6 months follow up and 12 months follow up measured by Psychological Assessment Tool 2.0 (PAT2.0) and Family Impact Module 2.0 (FIM2.0) in the intervention group versus the control group.
Siblings perception measured by the Siblings Perception Questionnaire (SPQ) | Baseline, 6 months and 12 months
  A change in siblings' perception of how cancer affected their daily life from baseline to 6 months and 12 months follow-up measured by Sibling Perception Questionnaire (SPQ) in the intervention group versus the control group.
Quality of life measured by Pediatric Quality of Life (PedsQL) | Baseline, 6 months and 12 months
  An enhancement in quality of life in childhood cancer survivors, their siblings and parents from baseline to 6 month and 12 month follow-up measured by Pediatric Quality of Life (PedsQL) in the intervention group versus the control group
Self reported sick leave in parents | Baseline, 6 months and 12 months
  A larger reduction in sick leave for parents from baseline to 6 month and 12 month follow-up measured by self reporting in the intervention group versus the control group.
Less stress induced telomere shortening | Baseline and 12 months
  A 10 ml blood sample to measure whether a psychosocial intervention results in a less shortening of the telomere length amongst parents of childhood cancer survivors from baseline to 12 months follow up versus parents in the control group
Anxiety and depression in parents of childhood cancer survivors measured by the Symptom Checklist (SCL) | Baseline, 6 months and 12 months
  A larger reduction in anxiety and depression symptoms in parents of childhood cancer survivors in the intervention group from baseline to 6 and 12 months follow up compared to the control group
Anxiety and depression in siblings over 18 years of childhood cancer survivors measured by the Symptom Checklist (SCL) | Baseline, 6 months and 12 months
  A larger reduction in anxiety and depression symptoms in siblings over 18 years of childhood cancer survivors in the intervention group from baseline to 6 and 12 months follow up compared to the control group
Anxiety and depression in childhood cancer survivors and their siblings i the age range 8 to 17 years measured by the Revised Child Anxiety and Depression Scale (RCADS) | Baseline, 6 months and 12 months
  A larger reduction in anxiety and depression symptoms in childhood cancer survivors and their siblings i the age range 8 to 17 years in the intervention group from baseline to 6 and 12 months follow up compared to the control group

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Johansen, Phd, Dr. MEd, Principal Investigator — Danish Cancer Society; Hanin Salem, Phd student, Principal Investigator — Danish Cancer Society
Locations (1):
- Danish Cancer Society, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bidstrup PE, Salem H, Andersen EW, Schmiegelow K, Rosthoj S, Wehner PS, Hasle H, Dalton SO, Johansen C, Kazak AE. Effects on Pediatric Cancer Survivors: The FAMily-Oriented Support (FAMOS) Randomized Controlled Trial. J Pediatr Psychol. 2023 Jan 12;48(1):29-38. doi: 10.1093/jpepsy/jsac062. PMID 35849020
- [Derived] Salem H, Kazak AE, Andersen EW, Belmonte F, Johansen C, Schmiegelow K, Winther JF, Wehner PS, Hasle H, Rosthoj S, Bidstrup PE. Home-based cognitive behavioural therapy for families of young children with cancer (FAMOS): A nationwide randomised controlled trial. Pediatr Blood Cancer. 2021 Mar;68(3):e28853. doi: 10.1002/pbc.28853. Epub 2020 Dec 27. PMID 33369038